CLINICAL TRIAL: NCT02652104
Title: A Review of the Clinical Outcome of Deep Brain Stimulation in the Patients With Advanced Parkinson's Disease in Helsinki and Uusimaa Hospital Between 2006 to 2014
Brief Title: Deep Brain Stimulation in HUCH Region Between 2006 and 2014
Status: Completed | Type: Observational
Sponsor: Hospital District of Helsinki and Uusimaa (Other)
Responsible Party: Principal Investigator, Maija Koivu, specialising physician, Hospital District of Helsinki and Uusimaa
Other Study IDs: Helsinki University Hospital
Record Dates: First submitted 2015-09-27; First posted 2016-01-11 (Estimated); Last update posted 2016-01-11 (Estimated); Status verified 2016-01

CONDITIONS: Parkinson's Disease
Keywords: Advanced; Deep brain stimulation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Only
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study reviews the outcome of deep brain stimulation treated patients in Helsinki and Uusimaa University Hospital between 2006 and 2014. The aim of the study is to investigate the outcome and possible side effects of deep brain stimulation treatment.

DETAILED DESCRIPTION:
Deep brain stimulation is a FDA approved method in treating patients with advanced Parkinson's disease when the best medical treatment is insufficient. In this study the aim is to investigate the outcome of deep brain stimulation treated patients in Helsinki and Uusimaa University hospital between 2006 and 2014. This study is a retrospective study based on existing patients' medical records and does not include an intervention in the treatment of an individual patient.

Deep brain stimulation carries the risks of major surgery. A complication risk for a hemorrhage is 1-2 % and for an infection is 3-10%. The aim of this study is to evaluate the complications that have occurred and the possible benefit of deep brain stimulation in deep brain stimulation treated patients with advanced Parkinson's disease.

The gathered data will be processed anonymously and an individual patient cannot be identified. The data will be processed with an appropriate statistical program (SPSS). No data will be given to external parties.

ELIGIBILITY:
Inclusion Criteria:

* Patient with advanced Parkinson's disease and given deep brain stimulation according to the best clinical protocol. This study only observes the outcome of given deep brain stimulation and does not affect on the given treatment.

Exclusion Criteria:

* The normal exclusion criteria for deep brain stimulation which are dementia, a significant vascular atrophy seen in brain CAT scan or MRI, Parkinson's disease with non-levodopa response with less than 30 % improvement in levodopa challenge test, disease duration less than 5 years

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consist of the patients who have received deep brain stimulation treatment. The patient selection for deep brain stimulation has been done according to a clinical protocol.
Sampling Method: Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2006-01; Primary Completion 2014-12 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
The benefit of deep brain stimulation in the well-being (measured in UPDRS III, H&Y scale) of a patient with advanced Parkinson's disease | at six months post-DBS

SECONDARY OUTCOMES:
The possible complications of deep brain stimulation in patient with advanced Parkinson's disease | years
The possible decrease in dosage of anti-Parkinsonian drugs after deep brain stimulation | years

CONTACTS AND LOCATIONS:
Overall Officials: Eero Pekkonen, M.D.,Ph.D., Study Director — Chief Physician